CLINICAL TRIAL: NCT01134796
Title: Assessment of GRASP II Medical Device to Improve Arm Coordination After Stroke
Brief Title: Assessment of GRASP Medical Device to Improve Arm Coordination After Stroke
Status: Terminated | Type: Observational
Why Stopped: failure to recruit
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 09103
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assessment of a custom made grasp device in the rehabilitation of stroke victims.

ELIGIBILITY:
Inclusion Criteria:

1. Damage to the following areas of the brain, all of which may be involved in coordination of reach to grasp confirmed by CT scan: parietal, cerebellar, internal capsule and basal ganglia,
2. A score of 6 or more on the arm section of the Rivermead Motor Assessment (able to reach and pick up a tennis ball and release on thigh),
3. Time between start of hand opening and start of hand transport > 60 ms (measured with GRASP).

Exclusion Criteria:

1. Cognitive dysfunction which prevents understanding of the task,
2. Severe concurrent medical problems that prevent repetitive reaching (including shoulder pain),
3. A diagnosis of Parkinson's disease, or
4. Lack of informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Stroke pateints and healthy volunteers (controls)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time to grasp | 3 sessions
  Primary outcome measures are: 1) The time elapsed between the start of grasp (when the finger breaks contact with the thumb) and the start of transport (when the wrist leaves the start position); and 2) The time elapsed between maximum aperture of the hand and peak deceleration of the wrist. Secondary outcome measures are: 1) movement duration, 2) time of maximum aperture expressed as % of movement duration, 3) time of peak deceleration expressed as % of movement duration, 4) amplitude of peak velocity of the wrist, 5) time of peak velocity, 6) time of peak velocity of the wrist expressed as % movement duration, 7) size of maximum aperture, 8) time to close hand from time of maximum aperture, 9) distance to target at time of maximum aperture.

CONTACTS AND LOCATIONS:
Overall Officials: Paulette Van Vliet, Principal Investigator — University of Nottingham